CLINICAL TRIAL: NCT06399159
Title: An Interpretable Multimodal Model Based on Cytology Ultrasound Noninvasively Predicts Lymph Node Metastasis in cN0 Papillary Thyroid Cancer
Brief Title: Prediction of Cervical Lymph Node Metastasis in Papillary Thyroid Carcinoma Based on Ultrasound and Cytological Images
Status: Completed | Type: Observational
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Xiachuan Qin,MD, Professor, Nanchong Central Hospital
Other Study IDs: Review-2023-109
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Papillary Thyroid Carcinoma; Lymph Node Metastasis
Keywords: ultrasound; deep learning; cytology
MeSH Terms: conditions — Thyroid Cancer, Papillary; Lymphatic Metastasis | interventions — Thyroidectomy; Lymph Node Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort with Lymph Node Metastasis: Depending on the pathological findings, it is classified as the presence of lymph node metastases.
  Interventions: Procedure: Thyroidectomy and lymph node dissection
- Cohort without Lymph Node Metastasis: Depending on the pathological findings, it is classified as the absence of lymph node metastases.
  Interventions: Procedure: Thyroidectomy and lymph node dissection

INTERVENTIONS:
Procedure: Thyroidectomy and lymph node dissection — All surgical specimens of thyroidectomy and lymph node dissection were subjected to paraffin-embedded histopathological examination, and postoperative were categorized as with cervical lymph node metastasis and without cervical lymph node metastasis.

SUMMARY:
Rising thyroid carcinoma rates, with papillary thyroid carcinoma (PTC) as the main type (85-90% of cases), often show early cervical lymph node spread. This increases the risk of PTC patients for recurrence and death. A new study's multimodal model fuses preoperative US and cytology images to better predict lymph node metastasis, aiming to improve treatment plans, reduce unnecessary surgeries, and enhance patient outcomes.

DETAILED DESCRIPTION:
Thyroid carcinoma incidence has been on the rise in recent years. Papillary thyroid carcinoma is the most prevalent type of differentiated thyroid carcinoma, accounting for 85% to 90% of malignant thyroid tumors. Despite its indolent nature, cervical lymph node metastasis is frequently observed at an early stage. Papillary thyroid carcinoma patients with cervical lymph node metastasis face an elevated risk of recurrence, distant metastasis, and mortality. Thus, non-invasive preoperative prediction of cervical lymph node metastasis is particularly vital for guiding treatment plans and prognostic. this study has developed a multimodal model integrating preoperative US images with cytological images of papillary thyroid carcinoma patients. The aim is to enhance the predictive accuracy for cervical lymph node metastasis, reduce unnecessary lymph node dissections, and provide real-time, precise guidance for determining the extent of surgical resection and prognostic assessment. This approach aims to optimize patient treatment strategies and enhance therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Underwent thyroidectomy and bilateral lymph node dissection with pathological confirmation of PTC
* Completed US examination within one week before surgery
* Underwent preoperative us-guided FNAC
* Completed cytological images at 400× magnification under a microscope

Exclusion Criteria:

* Patients who underwent only unilateral thyroidectomy
* Patients with cervical lymph nodes shown on preoperative ultrasound

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with papillary thyroid cancer from ten hospitals in China
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of lymph node metastasis | October 2024
  All surgical specimens were subjected to paraffin-embedded histopathological examination，depending on the pathological findings, it is classified as the presence or absence of lymph node metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Xiachuan Qin, MD, Study Chair — Nanchong Central Hospital
Locations (1):
- Nanchong central hospital, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided